CLINICAL TRIAL: NCT01515293
Title: Prospective Randomised Study Comparing Single Incision Transumbilical Versus Conventional Laparoscopic Appendectomy
Brief Title: Single Incision Versus Conventional Laparoscopic Appendectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Dolores Frutos Bernal, Dolores Frutos HUV Arrixaca, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUV-APP-MDFB
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2011-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Incision Laparoscopic Appendectomy (Experimental)
  Interventions: Procedure: Single Incision Laparoscopic Appendectomy
- Conventional appendectomy (Experimental): Conventional appendectomy
  Interventions: Procedure: Conventional appendectomy

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Appendectomy
  Arms: Single Incision Laparoscopic Appendectomy
Procedure: Conventional appendectomy
  Arms: Conventional appendectomy

SUMMARY:
The aim of this study is to compare the short-term outcomes of single-incision and conventional laparoscopic appendectomy.

DETAILED DESCRIPTION:
Appendicitis is the most common abdominal emergency. The treatment is surgical and single incision laparoscopic surgery (SILS) involves performing laparoscopic surgery through a single transumbilical point, in an attempt to improve the results of laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute appendicitis

Exclusion Criteria:

* Perforated appendicitis

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual)

REFERENCES:
- [Derived] Frutos MD, Abrisqueta J, Lujan J, Abellan I, Parrilla P. Randomized prospective study to compare laparoscopic appendectomy versus umbilical single-incision appendectomy. Ann Surg. 2013 Mar;257(3):413-8. doi: 10.1097/SLA.0b013e318278d225. PMID 23386239